CLINICAL TRIAL: NCT02709499
Title: Effects of the Low-level Laser Therapy on Inflammatory Profile on Patients With Coronary Artery Bypass Surgery: A Randomized, Controlled Clinical Trail
Brief Title: Effects of the Low-level Laser Therapy on Inflammatory Profile of the Patients With Coronary Artery Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, Clinical Research, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLLT-CABG-2016/2
Record Dates: First submitted 2016-02-18; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0J LLLT (Sham Comparator): The intervention will be made with the machine off.
  Interventions: Device: 0J LLLT
- 6J LLLT (Experimental): The Laser radiation will be made with 4J by spot
  Interventions: Device: 6J LLLT

INTERVENTIONS:
Device: 0J LLLT — perform with the machine off
  Other Names: Sham Low-Level Laser Therapy (Sham LLLT)
  Arms: 0J LLLT
Device: 6J LLLT — irradiation will be perform with 4J
  Other Names: 4J Low-Level Laser Therapy (4J LLLT)
  Arms: 6J LLLT

SUMMARY:
Cardiovascular diseases are the leading causes of morbidity and mortality in Brazil and surgical procedures to treat these disorders have grown dramatically in recent years. Since the first heart surgery in successful open field in humans, conducted in 1953 by John Lewis, many techniques have been used to improve the outcome of surgery and reduce their side effects. The low-level laser therapy (LBP) has been widely used in clinical practice for pain relief purposes, reducing inflammation and stimulating tissue healing. However, the effect of this therapy has been little elucidated in patients with cardiac disease. The objective of this study is to evaluate the effect of low level laser therapy on the inflammatory profile and cardiac tissue healing markers of patients in the postoperative period of CABG surgery.

DETAILED DESCRIPTION:
This study will be conducing in a large hospital that is reference in Cardiovascular diseases treatments. 38 patients will be randomized for placebo or 6J low-level laser therapy (LLLT). The inflammatory profile and cardiac tissue will be assessment before and after de LLLT.

ELIGIBILITY:
Inclusion Criteria:

* Patients after elective coronary artery bypass surgery, hemodynamically stable, without ischemic changes and / or complex arrhythmias on the electrocardiogram, between 45 and 75 years of age, who have performed the first surgery

Exclusion Criteria:

* Patients with decompensated heart failure; other associated surgery; presence of any comorbidity such as: unstable angina; sequel of stroke; photosensitivity; use of cardiac pacemaker; Diabetes mellitus (due to the negative effect of diabetes on wound healing).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
cytokine IL-10 | six days
cytokine IL-6 | six days
cytokine TNF-α | six days

SECONDARY OUTCOMES:
Troponin | six days
Creatine phosphokinase (CK) | six days
Lactate dehydrogenase (LDH) | six days
Complete blood count | six days
Visual Analog scale | six days
Hospital stay | six days
Pulmonary complications | six days

IPD SHARING:
Plan to Share IPD: No